CLINICAL TRIAL: NCT06632990
Title: An Open-label, Randomized, Three-arm Study Evaluating the Potential of BMS-984923 to Alter the Systemic Exposure of Three Orally Administered Probe Substrates in Healthy Adult Participants
Brief Title: A Study Evaluating the Potential of BMS-984923 to Alter the Systemic Exposure of Three Orally Administered Probe Substrates
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Allyx Therapeutics (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ALX-923-108; SB1AG087748 (NIH)
Record Dates: First submitted 2024-09-30; First posted 2024-10-09 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Drug Drug Interaction (DDI)
Keywords: Alzheimer's Disease; Synapses; Cognition; Neuroprotection; Neurons; mGluR5; metabolism
MeSH Terms: interventions — Midazolam; Caffeine; Dextromethorphan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 50 mg Active once daily (Experimental)
  Interventions: Drug: BMS-984923
- 50 mg Active twice daily (Experimental)
  Interventions: Drug: BMS-984923
- 100 mg Active twice daily (Experimental)
  Interventions: Drug: BMS-984923
- Reference drugs cocktail (Experimental): midazolam, caffeine and dextromethorphan will be administered orally
  Interventions: Drug: Midazolam; Drug: Caffeine; Drug: dextromethorphan

INTERVENTIONS:
Drug: BMS-984923 — oral capsules once or twice daily
  Other Names: ALX-001
  Arms: 100 mg Active twice daily; 50 mg Active once daily; 50 mg Active twice daily
Drug: Midazolam — midazolam, oral, 2mg administered before study drug and after study drug
  Arms: Reference drugs cocktail
Drug: Caffeine — Caffeine, oral, 100mg administered before study drug and after study drug
  Arms: Reference drugs cocktail
Drug: dextromethorphan — dextromethorphan, oral, 30mg administered before study drug and after study drug
  Arms: Reference drugs cocktail

SUMMARY:
The goal of this study is to learn if the investigational drug, BMS-984923 will impact the exposure and clearance of other medications when given together. Most drugs are broken down and cleared in the body via cytochrome P450 enzymes in the liver. The metabolism and clearance of certain drugs can be affected by other drugs when dosed together. To evaluate the impact of BMS-984923 on the clearance of other medications, we will investigate three known pathways which may be impacted by BMS-984923.

In this study participants will take one dose of the three known medications, midazolam, caffeine and dextromethorphan together. These drugs are known to be cleared by different cytochrome P450 enzymes. Blood will be collected to evaluate the exposure and clearance of these medications and their primary metabolites. Study participants will then be administered BMS-984923 for 18-days. On the 18th Day of BMS-984923 dosing, participants will again be co-administering midazolam, caffeine and dextromethorphan. Blood will be collected again, and the concentration of each drug will be measured. We will learn in this study if BMS-984923 changes the exposure and metabolism of the known drugs. These results will inform how BMS-984923 can be administered to patients who take multiple medications.

DETAILED DESCRIPTION:
To expand the use of concomitant medications in the future, the Sponsor is performing the clinical trial ALX-923-108 to determine the net effect (inhibition and induction) of BMS-984923 repeat dosing at 3 different clinically relevant doses of BMS-984923 on the pharmacokinetics of the sensitive cytochrome P450 probe substrates caffeine (CYP1A2), dextromethorphan (CYP2D6), and midazolam (CYP3A4) and their respective metabolites as measured by systemic exposure of each probe.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between the ages of 18 and 50 years, inclusive.
* No history of cognitive impairment.
* Capable of providing written informed consent and willing to comply with all study requirements and procedures.
* Female participants, if of childbearing potential, must be non-lactating, confirmed to be non-pregnant (negative serum pregnancy test), and agree to use a highly effective form of contraception throughout the trial and for 90 days after the last dose.
* Male participants who are sexually active with a woman of childbearing potential must agree to use condoms during the study and for 90 days after the last dose unless the woman is using a highly effective form of contraception
* Compliance with restricted foods, medications, and drinks outlined within this protocol

Exclusion Criteria:

* Currently on any medication for a chronic condition.
* Any significant neurologic disease, such as AD, Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.
* A current DSM V diagnosis of active major depression, schizophrenia, or bipolar disorder.
* Positive urine drug screen or positive urine alcohol or alcohol breathalyzer test.
* Current use of cannabidiol / THC.
* Current nicotine use or positive urine cotinine test.
* Participants must test negative for caffeine prior to dosing.
* History of alcohol or substance abuse or dependence within the past 2 years (DSM-IV criteria).
* Clinically significant or unstable medical condition, including uncontrolled hypertension, uncontrolled diabetes, or significant cardiac, pulmonary, renal, hepatic, endocrine, or other systemic disease that, in the opinion of the PI, may either put the participant at risk because of participation in the study, or influence the results, or the participant's ability to participate in the study.
* Any disorder or medication that could interfere with the absorption, distribution, metabolism or excretion of drugs (e.g., small bowel disease, Crohn's disease, celiac disease, GERD, or liver disease and antimotility or gastric acid depressing medications and weight loss medications)
* Surgical history of the GI tract affecting gastric motility or altering the GI tract (with the exception of uncomplicated appendectomy and hernia repair) (a cholecystectomy is exclusionary).
* Use of medications with potential drug-drug interactions
* Is unable to refrain from the use of other prescription or non-prescription drugs
* History or presence of clinically significant ECG abnormalities
* Donation of blood or blood products for transfusion within 3 months prior to first study drug administration
* History of hypersensitivity to any of the excipients in the formulation of the study drugs.
* History of hypersensitivity to midazolam, caffeine, or dextromethorphan or any other formulation ingredients.
* Use of another investigational agent within 30 days or 5 half-lives
* Neutropenia
* Thrombocytopenia
* Has moderate or severe renal disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-04-03 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Area under the curve for the first and last 96 hours of dosing (AUC96h) as determined by PK modeling | 24 days
  Total plasma concentration of caffeine as determined by pharmacokinetic modeling
Area under the curve for the first and last 96 hours of dosing (AUC96h) as determined by PK modeling | 24 days
  Total plasma concentration of midazolam as determined by pharmacokinetic modeling
Area under the curve for the first and last 96 hours of dosing (AUC96h) as determined by PK modeling | 24 days
  Total plasma concentration of dextromethorphan as determined by pharmacokinetic modeling
Area under the curve for the last 96 hours of dosing (AUC96h) | last 96 hours
  Total plasma concentration of BMS-984923 as determined by pharmacokinetic modeling
Trough plasma drug concentration at steady state | 21 days
  plasma concentration of BMS-984923 as determined by pharmacokinetic modeling

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) Safety | 30 days
  Safety
Incidence of clinically significant lab abnormalities | 30 days
  Safety
Incidence of clinically significant changes in safety assessments vital signs, physical exam, electrocardiogram | 30 days
  Safety

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No